CLINICAL TRIAL: NCT00014066
Title: A Phase I Study of Photodynamic Therapy (PDT) Combined With High Dose Rate (HDR) Brachytherapy for Patients With Obstructive Bronchogenic Carcinoma
Brief Title: Photodynamic Therapy Plus Brachytherapy in Treating Patients With Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Purpose: Treatment
Other Study IDs: DS 92-40; RPCI-DS-92-40; NCI-V97-1190
Record Dates: First submitted 2001-04-10; First posted 2004-02-04 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; recurrent non-small cell lung cancer; limited stage small cell lung cancer; recurrent small cell lung cancer; stage 0 non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Hematoporphyrin Derivative; Brachytherapy

INTERVENTIONS:
Drug: hematoporphyrin derivative
Radiation: brachytherapy

SUMMARY:
RATIONALE: Photodynamic therapy uses light and drugs that make cnacer cells more sensitive to light to kill tumor cells. Brachytherapy uses radiation to damage tumor cells. Photodynamic therapy combined with brachytherapy may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of photodynamic therapy plus brachytherapy in treating patients with recurrent lung cancer that is blocking the lung passages.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the feasibility, toxicity, and effectiveness of combination therapy with Photofrin PDT and HDT brachytherapy in patients with endobronchial obstructions from lung cancer.

OUTLINE: This is not a randomized study. Photofrin solution is administered slowly as a bolus injection over 3-5 minutes on day 1. Bronchoscopy is performed under general anesthesia 48 hours after Photofrin injection. Light is transmitted from the laser to the tumor via quartz fiber optics (interstitial or surface PDT). Another bronchoscopy is performed 48 hours after PDT treatment to clean out any tissue debris left after PDT treatment. HDR brachytherapy is performed using prescribed dose of radiation for 5-10 minutes to designated positions. Repeat bronchoscopy is performed 3-4 weeks post HDR brachytherapy and a second HDR brachytherapy treatment may be given. Patients are followed every 3 months until death, or for 5 years.

PROJECTED ACCRUAL: 16 patients will be entered over 1.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed small cell or non-small cell primary lung cancer with symptomatic endobronchial lesion(s) partially or totally obstructing airway distal to the carina and accessible by endoscopy Recurrent disease following prior therapy and/or be ineligible for, or refuse, alternative standard therapy such as: Surgery External radiation therapy Chemotherapy High grade obstruction necessitating more rapid aeration and palliation than standard therapy can provide No evidence of encasement or extension of the tumor to the right or left major pulmonary vessels on CT of the chest No tumor involvement at trachea or carina

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: WBC at least 4,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 2 times the upper limit of normal SGOT/SGPT less than 2 times the upper limit of normal Renal: Creatinine no greater than 2.0 mg/dL Other: Not pregnant Adequate method of contraception required of all fertile patients Female fertile patients must have normal serum beta HCG Not eligible for standard therapy and/or other protocol therapy No hypersensitivity to DHE or other porphyrins Not concurrent photosensitizing drugs such as: Tetracycline Doxorubicin No contraindications to general anesthesia, including EKG abnormalities suggestive of acute ischemia

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No chemotherapy within 3 weeks prior to study entry No doxorubicin within 8 weeks prior to study entry Endocrine therapy: Not specified Radiotherapy: Prior radiation therapy dose no higher than 75 Gy to proposed bronchial segment allowed No concurrent external brain radiation therapy Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1993-03; Primary Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory M. Loewen, DO, FCCP, Study Chair — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States